CLINICAL TRIAL: NCT04963218
Title: A Multicenter Study of Detection of Low Ventricular Ejection Fraction (LVEF) ≤ 40% Based on Point-of-Care 12- Lead ECG Data
Brief Title: A Multi-Center Study of Detection of Low Ventricular Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Anumana, Inc. (Industry)
Responsible Party: Principal Investigator, Peter A. Noseworthy, M.D., Professor of Medicine, Mayo Clinic
Other Study IDs: 21-003530
Record Dates: First submitted 2021-07-01; First posted 2021-07-15 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AI Algorithm to detect LVEF in ECG — A clinical decision support software as a medical device that detects whether a patient has LVEF less than or equal to 40% based upon the input of one or more ECG vectors at the point-of-care.

SUMMARY:
This is a multi-site, retrospective study to evaluate the performance of a locked AI-based algorithm for detection of left ventricular systolic dysfunction. A prerequisite for inclusion of subjects from each institution will be the availability of at least one digital 12-lead ECG paired with an echocardiogram with LVEF information within 30 days of the date of the ECG. The AI-ECG LVSD algorithm will be applied on all ECGs and diagnostic performance features for the detection of LVSD will be estimated using the provided paired LVEF value (Low LVEF as the reference label). Performance will also be assessed in subgroups of subjects determined by demographic and clinical factors.

DETAILED DESCRIPTION:
Following institutional review board approval, 12,000 12-lead ECG's paired with an echocardiogram with LVEF information within 30 days of the date of the ECG will be collected across three enrolled sites. Each site will provide data from up to 4000 enrolled subjects that meet the inclusion criteria. No other demographic characteristics or enrichment will be considered in the selection of subjects in order to best represent the general population for that site. Sites will securely transfer the data to a centralized repository for processing.

Once data is collected, the device will be used to analyze the ECG data for all enrolled subjects without reference or access to the echocardiogram data. The device will display a binary 36 prediction of the likelihood of LVEF less than or equal to 40%. Results will be compared to the echocardiogram reference standard in accordance with the statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

- Adult subjects with or without known cardiac disease who are either inpatients or outpatients with ECGs and an echocardiogram within 30-days of the ECG date.

Exclusion Criteria:

* No research authorization provided
* An ECG signal shorter than 10 seconds or that is not interpretable
* An echocardiogram is considered technically challenging
* Only qualitative interpretation of left ventricular systolic function available (i.e., "decreased EF") without a numerical value.
* A paced rhythm

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with or without known cardiac disease who are either inpatients or outpatients with ECGs and an echocardiogram within 30-days of the ECG date.
Sampling Method: Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Established Diagnostic Performance | 1 month
  Number of participants with presence of EF less than of equal to 40% identified by 12-lead AI ECG algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Peter Noseworthy, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Beth Israel Deacon Medical Center, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Monument Health, Rapid City, South Dakota
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials